CLINICAL TRIAL: NCT03538600
Title: Sample Collection From Healthy Volunteers for Assay Optimization
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180101; 18-I-0101
Record Dates: First submitted 2018-05-25; First posted 2018-05-29 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11-24

CONDITIONS: Healthy Volunteers
Keywords: Blood; Microbiome Analysis; Stool; Saliva; Skin; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: healthy volunteers

SUMMARY:
Background:

The Laboratory of Immune System Biology (LISB) works with other labs at the National Institutes of Health. They study how parts of living things come together to make a whole. LISB designs and improves research tests on human samples like blood and cells. In order to do its work, LISB needs to have a lot of these samples available.

Objective:

To collect biological specimens to use for designing and improving research tests. Specimens include blood, stool, saliva, and skin/mucosal swabs.

Eligibility:

Healthy people ages 3-80

Design:

Participants will be screened with an interview about their general health and their medical history. They will have a physical exam and blood tests.

If the results of the screening are normal, participants will be asked to give one or more of these samples:

Blood will be drawn from an arm vein with a needle and syringe.

Mucus and skin will be collected by rubbing the area with a cotton swab. The areas may include the top of the tongue, inside the cheek, nostrils, behind the ear, elbow pit, or vagina.

Participants will spit into a tube to collect saliva.

Participants will pass stool into a plastic container that fits in the toilet under the seat. They will get sampling kits and instructions.

Over the next 5 years, if more samples are needed, participants will be contacted to set up another visit to the NIH. These visits will each take about 1 hour.

About every 2 years, when participants come to NIH for a visit, extra blood will be collected. It will be tested for HIV and hepatitis B and C.

DETAILED DESCRIPTION:
The Laboratory of Immune System Biology plays a major role in fostering the growth of systems biology efforts across the National Institutes of Health, in large measure through its development of new tools for high-throughput data generation and complex systems modeling. The lab s experimental component requires ongoing assay development and optimization, which depend on the availability of human biological samples for testing. The primary purpose of this protocol is to obtain biological specimens from healthy volunteers to support the lab s development and optimization of scientific assays, and to use as control samples for research tests in other studies. The secondary objective of this study is to track immunologic changes over time using the assays developed and optimized in this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Aged 3-80 years.
  2. Able to provide informed consent (for ages >=18 years) or has a parent or guardian who can provide informed consent on their behalf (for ages <18 years).
  3. Agree to allow biological samples to be stored for future research.
  4. Willing to provide blood, stool, saliva, skin/mucosal/tonsil swabs, and/or skin punch biopsy specimens.

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

1. Pregnancy.
2. History of autoimmune or autoinflammatory disease.
3. Diabetes mellitus.
4. Cancer chemotherapy within the past 5 years.
5. Currently receiving treatment for an active malignancy.
6. Surgery within the past 8 weeks.
7. History of recent (within the past 30 days) infection.
8. History of significant, active parasitic, amebic, fungal, or mycobacterial infections within the past 5 years (as determined by the PI).
9. Infected with HIV and/or hepatitis B and/or C.
10. Use of an oral or inhaled glucocorticoid within the past 30 days.
11. History of a bleeding disorder.
12. Screening lab values are both outside of the NIH Department of Laboratory Medicine normal reference range and deemed clinically significant by the PI.
13. Receipt of an immunosuppressant or immunomodulatory drug within the past 30 days.
14. Receipt of a live-attenuated vaccine within the past 30 days.
15. Receipt of any other type of vaccine within the past 14 days.
16. Current or past use (within the past 90 days) of immunoglobulin therapy.
17. Current use of illicit drugs (per subject report).
18. Current use of nicotine-containing products, including cigarettes and chewing tobacco, nicotine patches, gum, electronic cigarettes, etc.
19. Current alcohol use disorders (criteria per Diagnostic and Statistical Manual of Mental Disorders, fifth edition).
20. Any condition that requires active medical intervention or monitoring to avert serious danger to the individual s health or wellbeing.
21. Any condition that, in the opinion of the PI, contraindicates participation in this study or would significantly affect immune profile.

Co-enrollment guidelines: Participants may be co-enrolled in other studies. The PI may withdraw them from this study for any reason that may contraindicate participation.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy Volunteers between the ages of 3-80.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-06-28 (Actual); Primary Completion 2043-06-30 (Estimated); Study Completion 2043-06-30 (Estimated)

PRIMARY OUTCOMES:
The purpose of this study is to collect biological specimens (blood, stool, saliva, skin/mucosal swabs, and/or skin punch biopsy specimens) for the development and optimization of scientific assays, and to use as control samples for research tes... | Throughout the study.
  The purpose of this study is to collect biological specimens (blood, stool, saliva, skin/mucosal swabs, and/or skin punch biopsy specimens) for the development and optimization of scientific assays, and to use as control samples for research tests in other studies.. There is no specified outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kalpana Manthiram, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-I-0101.html